CLINICAL TRIAL: NCT05669196
Title: Evaluation of Respiratory Muscle Strength, Diaphragmatic Thickness and Functional Exercise Capacity in Lobectomy Surgeries With Thoracotomy and VATS
Brief Title: Diaphragmatic Thickness and Functional Exercise Capacity in Lobectomy Surgeries With Thoracotomy and VATS
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Funda Sirakaya, Doctorate student, Hacettepe University
Other Study IDs: KA-19084
Record Dates: First submitted 2022-10-19; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-11

CONDITIONS: Video Assisted Thoracoscopic Surgery; Thoracic Surgery; Respiratory Muscles
Keywords: Lung cancer, functional capacity
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- standard thoracotomy group: Individuals who are between the ages of 18-75 and lung cancer patient, underwent lobectomy with standard thoracotomy
- muscle sparing thoracotomy group: Individuals who are between the ages of 18-75 and lung cancer patient, underwent lobectomy with muscle sparing thoracotomy
- VATS group: Individuals who are between the ages of 18-75 and lung cancer patient, underwent lobectomy with video-assisted thoracic surgery

SUMMARY:
The most commonly treatment for early stage non-small cell lung cancer (NSCLC) is lobectomy. Different surgical interventions during lobectomy are thought to have different effects on respiratory functions and exercise capacities. The aim of this study was to evaluate respiratory muscle strength, functional exercise capacity, and diaphragmatic thickness in groups that underwent lobectomy with standard thoracotomy, muscle sparing thoracotomy, and video-assisted thoracic surgery (VATS).

DETAILED DESCRIPTION:
The most commonly treatment for early stage non-small cell lung cancer (NSCLC) is lobectomy. Different surgical interventions during lobectomy are thought to have different effects on respiratory functions and exercise capacities. The aim of this study was to evaluate respiratory muscle strength, functional exercise capacity, and diaphragmatic thickness in groups that underwent lobectomy with standard thoracotomy, muscle sparing thoracotomy, and video-assisted thoracic surgery (VATS). In this study we will evaluate respiratory muscle strength, functional exercise capacity, diaphragmatic thickness, postoperative pulmonary complications, pain, dyspnea, pulmonary function, functional status, anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Being a lung cancer patient scheduled for standard thoracotomy, muscle sparing thoracotomy, or lobectomy with VATS,
* Being clinically stable,
* Volunteering to participate in the study,
* be between the ages of 18-75,
* To be cooperative in the tests to be done.

Exclusion Criteria:

* Having an orthopedic and neurological condition that prevents walking, - Having undergone any surgery on the thoracic wall,
* Diagnosed with small cell lung cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with lung cancer who met the inclusion criteria in the 18-75 age range participated in the study. According to the surgical intervention methods, the patients in our study; divided into three groups as standard thoracotomy, muscle sparing thoracotomy, and VATS.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength (inspiration) change | The day before the operation.
  Respiratory muscle strength will measure by measuring mouth pressure and using maximal inspiratory pressure (MIP) values. Preoperative and postoperative value differences will be calculated.
Respiratory muscle strength (inspiration) change | 15-20 days after discharge.
  Respiratory muscle strength will measure by measuring mouth pressure and using maximal inspiratory pressure (MIP) values. Preoperative and postoperative value differences will be calculated.
Respiratory muscle strength (expiration) change | The day before the operation.
  Respiratory muscle strength will measure by measuring mouth pressure and using maximal expiratory pressure (MEP) values. Preoperative and postoperative value differences will be calculated.
Respiratory muscle strength (expiration) change | 15-20 days after discharge.
  Respiratory muscle strength will measure by measuring mouth pressure and using maximal expiratory pressure (MEP) values. Preoperative and postoperative value differences will be calculated.

SECONDARY OUTCOMES:
Functional exercise capacity | The day before the operation.
  6-minute walk test (6MWT) will be used to evaluate functional exercise capacity.
Functional exercise capacity | 15-20 days after discharge.
  6-minute walk test (6MWT) will be used to evaluate functional exercise capacity.
Diaphragmatic thickness | The day before the operation.
  Ultrasound will be used to measure diaphragmatic thickness.
Diaphragmatic thickness | 15-20 days after discharge.
  Ultrasound will be used to measure diaphragmatic thickness.
Postoperative Pulmonary Complication | Postoperative first-fifth days.
  Postoperative pulmonary complications will be evaulate by Melbourne Group Scale. If more than 4 parameters are positive, it will be considered as having postoperative pulmonary complication.
Postoperative pain | The operative day after the operation.
  Visual anolog scala will be used to measure pain. Zero is considered as no pain an ten s considered as no maximal pain.
Postoperative pain | Postoperative first-fifth days.
  Visual anolog scala will be used to measure pain. Zero is considered as no pain an ten s considered as no maximal pain.
Postoperative pain | 15-20 days after discharge.
  Visual anolog scala will be used to measure pain. Zero is considered as no pain an ten s considered as no maximal pain.
Dyspnea | The day before the operation.
  Dyspnea will be evaulate by Modifiye Medical Research Council Dyspnea Scale (mMRC).
Dyspnea | 15-20 days after discharge.
  Dyspnea will be evaulate by Modifiye Medical Research Council Dyspnea Scale (mMRC).
Pulmonary function (FEV1) | The day before the operation.
  Pulmonary function will be evaulate by pulmonary function test. FEV1 will be measured in liter.
Pulmonary function (FEV1) | 15-20 days after discharge.
  Pulmonary function will be evaulate by pulmonary function test. FEV1 will be measured in liter.
Pulmonary function (FVC) | The day before the operation.
  Pulmonary function will be evaulate by pulmonary function test. FVC will be measured in liter.
Pulmonary function (FVC) | 15-20 days after discharge.
  Pulmonary function will be evaulate by pulmonary function test. FVC will be measured in liter.
Pulmonary function (FEF25-75) | The day before the operation.
  Pulmonary function will be evaulate by pulmonary function test. FEF25-75 will be measured in liter.
Pulmonary function (FEF25-75) | 15-20 days after discharge.
  Pulmonary function will be evaulate by pulmonary function test. FEF25-75 will be measured in liter.
Pulmonary function (PEF) | The day before the operation.
  Pulmonary function will be evaulate by pulmonary function test. PEF will be measured in liter.
Pulmonary function (PEF) | 15-20 days after discharge.
  Pulmonary function will be evaulate by pulmonary function test. PEF will be measured in liter.
Functional Status | The day before the operation.
  Karnofsky Performance Status Scale will be used to evaluate functional status. It will be used i to assess the preoperative condition.
Anxiety and Depression | Postoperative first-fifth days.
  Anxiety and depression will be evaulate by Hospital Anxiety and Depression Scale. 7 of the survey questions question depression and 7 of them question anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Sirakaya, MsC, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No